CLINICAL TRIAL: NCT01715220
Title: Treatment of Suspected Cholelithiasis With Nitroglycerin: a Randomized, Prospective Double-blind Trial
Brief Title: Treatment of Suspected Cholelithiasis With Nitroglycerin
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMCSD.2012.0003
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: COLIC; BILIARY TRACT DISEASES
Keywords: Nitroglycerin; Biliary Colic; Cholelithiasis; Abdominal Pain.
MeSH Terms: conditions — Colic; Biliary Tract Diseases; Cholelithiasis; Abdominal Pain | interventions — Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sublingual nitroglycerine (Active Comparator): Sublingual nitroglycerine followed by pain assessment and if necessary second dose of sublingual nitroglycerine
  Interventions: Drug: sublingual nitroglycerine
- placebo (Placebo Comparator): sublingual placebo followed by pain assessment and if necessary second dose of sublingual placebo
  Interventions: Drug: sublingual nitroglycerine

INTERVENTIONS:
Drug: sublingual nitroglycerine — A convenience sample of patients presenting to the Emergency Department will be randomized to receive either sublingual 0.4 mg doses of nitroglycerin or placebo. Pain prior to and at two minutes and five minutes after medication administration will be assessed using a visual analog scale. The medication will be either a 0.4 mg dose of nitroglycerin or a placebo. If pain is not completely relieved within five minutes, a second dose will be administered after blood pressure assessment. If the pain is not completely relieved after an additional two minute and five minute assessment or the pain returns, it will be treated in the standard manner at the discretion of the treating Emergency Physician
  Other Names: Nitrolingual

SUMMARY:
ABSTRACT: Sublingual nitroglycerin has been advocated for the treatment of acute pain from suspected symptomatic cholelithiasis. There is, however, no clinical studies that validate its use. This study is designed to evaluate the efficacy of nitroglycerine in relieving acute pain of suspected biliary tract origin.

Nitroglycerin is a potent smooth muscle relaxant used for biliary tract dilation during ERCP, (Chelly, J) and has been recommended for treatment of biliary colic based on anecdotal experience and small case reports. Nitroglycerin effect is a result of the nitric oxide component of the medication which acts as a smooth muscle relaxant in vascular, bronchial, esophageal and biliary smooth muscles. [McGowan(1936), Chelly (1979),Toyoyama (2001)] The typical dose of nitroglycerin is 0.4 mg given sublingually in pill form or, more recently, in a metered spray form. In a case series reported by Hassel (1993), positive response times ranged from 20 to 60 seconds with duration of action of two to twelve hours. Sublingual nitroglycerin is most commonly used for treatment of chest pain related to insufficient cardiac perfusion. It has also been noted to relieve the pain of esophageal spasms. Nitroglycerin has an excellent safety profile if used in patients with adequate pretreatment blood pressures. [Newberry (2005), Nitroglycerine (2011), Nitro (2011), Wolters (2009)] This study proposes to compare sublingual 0.4 mg doses of nitroglycerin to placebo for the initial treatment of acute pain from suspected symptomatic cholelithiasis

DETAILED DESCRIPTION:
General Approach: This study proposes to compare sublingual 0.4 mg doses of nitroglycerin to placebo for initial treatment for acute pain from suspected symptomatic cholelithiasis. Patients with right upper quadrant abdominal pain of less than 24 hour duration between ages 18 and 60 years of age will be offered treatment with sublingual nitroglycerin or placebo. Patients with obstructive hypertrophic cardiomyopathy, pronounced hypovolemia, STEMI or presumed cardiac chest pain, inferior myocardial infarction with right ventricular involvement, raised intracranial pressure, cardiac tamponade, and patients taking certain drugs for erectile dysfunction (phosphodiesterase inhibitors), pregnancy, or with a known allergy to nitroglycerin will be excluded from the study.

2. Methods: A convenience sample of patients presenting to the Emergency Department will be randomized to receive either sublingual 0.4 mg doses of nitroglycerin or placebo. Pain prior to and at two minutes and five minutes after medication administration will be assessed using a visual analog scale. The medication will be either a 0.4 mg dose of nitroglycerin or a placebo. If pain is not completely relieved within five minutes, a second dose will be administered after blood pressure assessment. If the pain is not completely relieved after an additional two minute and five minute assessment or the pain returns, it will be treated in the standard manner at the discretion of the treating Emergency Physician. Ancillary studies and other treatments will be at the discretion of the treating physician. The 0.4mg dose of nitro has been proven to be a safe and well tolerated dose when administered to our patient population in treatment of acute coronary syndrome or suspected angina. Our attending, resident, and nursing staff are very familiar with this dose, the potential side effects of the medication, and its administration procedure. Therefore, we believe that 0.4mg will be a optimal starting dose for enrollees in our study.

3. Retrovirology Research: None

4. Investigational Drugs/Devices/Biologics Research: None

5. Statistical Analysis: Demographic information, patient characteristics, assignment to experimental group, and visual analog pain scale data will be entered into a spreadsheet . Pain will be recorded per patients at 5 time points: 0, 2, 5, 7, and 10 minutes. Descriptive statistics will be presented in tables and graphs. Pain scale results will be analyzed by a two-way (2x5) repeated measures analysis of variance with interaction and post hoc multiple comparisons. The primary time pair to be tested will be the difference between treatment and placebo groups in pain reduction from 0 to 2 minutes. The planned sample size is 62, with 31 in the placebo group and 31 in the nitro group. The sample size was calculated with the aid of Dr Riffenburgh. He agrees with sample size suggested above.

6. Military Relevance / Operational Use, if any: Sublingual nitroglycerin is a standard AMAL list item for independent providers in most field and operational settings. Relief of biliary colic can significantly reduce the number of urgent medical evacuations for right upper quadrant pain. There is also no mental status degradation with the use of nitroglycerin, unlike the opioids commonly used to treat biliary colic.

ELIGIBILITY:
Inclusion Criteria: Patients with right upper quadrant abdominal pain of less than 24 hours' duration between ages 18 and 60 years of age will be offered treatment with sublingual nitroglycerin or placebo.

Exclusion Criteria: Patients with obstructive hypertrophic cardiomyopathy, pronounced hypovolemia, alcohol use in the last 8 hours, clinical intoxication, STEMI or presumed cardiac chest pain, inferior myocardial infarction with right ventricular involvement, raised intracranial pressure, cardiac tamponade and patients taking certain drugs for erectile dysfunction (phosphodiesterase inhibitors), pregnancy or with a known allergy to nitroglycerin will be excluded from the study. Patients unable to give consent will be excluded.

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
pain relief on visual analog scale | two and five minutes
  pain relief assesement at two and five minutes after medication or placebo with standard treatment if inadequate pain relief.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Portouw, MD, Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No